CLINICAL TRIAL: NCT07130123
Title: Removal of the Intubation Tube Under Positive Pressure With or Without Endotracheal Suctioning During Extubation in Intensive Care: a Prospective Randomised Controlled Trial
Brief Title: Endotracheal Suctionning During Positive Pressure Extubation in ICU
Acronym: INTENTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUO-2025-12
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mechanical Ventilation With Oral Intubation; Weaning Invasive Mechanical Ventilation; Oxygen Saturation Measurement; Rox Index; Extubation
Keywords: rox index; extubation; Suctionning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suctionning Extubation (experimental arm) (Experimental): Endotracheal suctioning during positive pressure extubation in mechanically ventilated adult patients in the intensive care unit.
  Interventions: Procedure: Suctionning extubation
- No Suctionning Extubation (control arm) (Sham Comparator): No endotracheal suctioning during positive pressure extubation in mechanically ventilated adult patients in the intensive care unit.
  Interventions: Procedure: No suctionning Extubation

INTERVENTIONS:
Procedure: Suctionning extubation — We will remove the intubation tube with endotracheal suctioning during the extubation procedure and maintain positive end expiratory pressure (PEEP) and pressure support. The PEEP level will be 10 cmH2O and the pressure support 7 cmH2O for 2 minutes prior to extubation. The vacuum level will be the maximum level (standard procedure in the unit), i.e. 450 mmHg. The closed-system suction probe is inserted up to the last mark corresponding to 40cm. The size of our closed system is identical for all patients, i.e. 14 french.
  Arms: Suctionning Extubation (experimental arm)
Procedure: No suctionning Extubation — In the control group, removal of the intubation tube during the extubation procedure is performed with PEEP maintained, without endotracheal suctioning. The PEEP level will be set at 10 cmH2O and the pressure at 7 cmH2O in the 2 minutes prior to extubation.
  Arms: No Suctionning Extubation (control arm)

SUMMARY:
The aim of this clinical trial is to evaluate endotracheal suctioning during positive pressure extubation in mechanically ventilated adult patients (over 18 years old) in the intensive care unit (ICU). The main question it aims to answer is whether the intervention improves the respiratory oxygenation index (ROX) three hours after extubation compared to no endotracheal suction during positive pressure extubation.

Participants will only need to be extubated by the nursing team in the ICU. Follow-up will consist of evaluating respiratory rate, pulse oximetry and inspired oxygen fraction for three hours following extubation.

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled trial. The aim of this study is to evaluate endotracheal suctioning during positive pressure extubation in mechanically ventilated adult patients (over 18 years old) in the intensive care unit (ICU). The main question it aims to answer is whether the intervention improves the respiratory oxygenation index (ROX) three hours after extubation compared to no endotracheal suction during positive pressure extubation.

Inclusion : Participants who meet eligibility criteria will be randomized into experimental arm (endotracheal suctioning during positive pressure extubation) or control arm (no endotracheal suction during positive pressure extubation).

Intervention and Follow-up : participants will only need to be extubated by the nursing team in the ICU. Follow-up will consist of evaluating respiratory rate, pulse oximetry and inspired oxygen fraction for three hours following extubation.

End of study : at the end of the study visit (28 days after extubation), vital status of participants will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Intubated for more than 48 hours
* Patient for whom extubation is prescribed by the patient's physician

Exclusion Criteria:

* Headboard restriction>30°.
* Decision to limit active treatment in advance of reintubation
* Protected person (under guardianship or curatorship)
* Person under court protection
* Persons deprived of liberty
* Persons not affiliated to a social security scheme
* Pregnant or breast-feeding woman
* No co-inclusion with a study whose period of interest is follow-up within 3 hours of extubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Respiratoy/oxygenation index (ROX index) | 3 hours after extubation
  Rox index will be assessed 3 hours after extubation by an investigator with no information about randomization (blind assessment)

SECONDARY OUTCOMES:
Mechanical ventilation weaning failure | During 7 days after extubation
  Weaning failure corresponds with death or new intabution
ROX index evolution | During 3 hours after extubation
  Rox index will be assessed 3 times after extubation in order to evaluate its evolution (blind assessment) :
  1. 30 minutes after extubation
  2. 1 hour after extubation
  3. 3 hour after extubation
Pneumonia after extubation | During 7 days after extubation
  Rate of hospital-acquired pneumonia confirmed by an investigator
Airway clearance technique | During 24 hours after extubation
  Use of any airway clearance technique after extubation :
  * nasotracheal suction
  * respiratory physiotherapy
  * bronchial fibroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Cécile FOSSAT, Principal Investigator — Centre Hospitalier Universitaire d'Orléans
Locations (1):
- Centre Hospitalier Universitaire d'Orléans, Orléans, Loiret, France

REFERENCES:
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Frutos-Vivar F, Esteban A, Apezteguia C, Gonzalez M, Arabi Y, Restrepo MI, Gordo F, Santos C, Alhashemi JA, Perez F, Penuelas O, Anzueto A. Outcome of reintubated patients after scheduled extubation. J Crit Care. 2011 Oct;26(5):502-509. doi: 10.1016/j.jcrc.2010.12.015. Epub 2011 Mar 3. PMID 21376523
- [Background] Fossat G, Desmalles E, Courtes L, Fossat C, Boulain T. Cough Peak Flow Assessment Without Disconnection From the ICU Ventilator in Mechanically Ventilated Patients. Respir Care. 2023 Apr;68(4):470-477. doi: 10.4187/respcare.10412. Epub 2023 Mar 6. PMID 36878644